CLINICAL TRIAL: NCT02500992
Title: Bacterial Contamination in Transrectal Hybrid Natural Orifice Translumenal Endoscopic Surgery Sigmoidectomy for Diverticular Disease
Brief Title: Bacterial Contamination in Transrectal Hybrid NOTES Sigmoidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Daniel Steinemann, MD, Consultant, Cantonal Hosptal, Baselland
Other Study IDs: NoBakt transrectal
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Diverticular Disease
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbacteriological swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transrectal sigmoidectomy: Patients undergoing transrectal NOTES sigmoidectomy
  Interventions: Procedure: Transrectal sigmoidectomy
- Laparoscopic-assisted sigmoidectomy: Patients undergoing laparoscopic-assisted sigmoidectomy

INTERVENTIONS:
Procedure: Transrectal sigmoidectomy
  Groups: Transrectal sigmoidectomy

SUMMARY:
Transrectal Hybrid natural orifice translumenal endoscopic surgery sigmoidectomy has gained popularity. It is an appealing technique as a minilaparotomy in order to retrieve the specimen is avoided. Therefore less postoperative pain and a better cosmetic result are expected. The feasibility of the technique has been demonstrated.

Still an open question is the risk of intraperitoneal contamination as in this procedure the colon has to be opened. This is the case for (a) retrieval of the specimen thru the opened rectal stump and (b) for intracorporeal insertion of the anvil of the circular stapler in order to fashion an anastomosis.

In this study the bacterial contamination in the rectal stump as well as in the peritoneal cavity is assessed. The results are compared to bacteriological samples taken in a comparison group consisting of conventional laparoscopic assisted sigmoidectomies.

ELIGIBILITY:
Inclusion Criteria:

* Status post several episodes of diverticulitis
* Status post contained diverticulitis

Exclusion Criteria:

* not able to give informed consent
* <18 years of age
* pregnancy
* emergency operation
* acute diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for elective sigmoidectomy for diverticular disease. Status post several episodes of diverticulitis, status post contained diverticulitis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Peritoneal bacterial contamination | during surgery
  microbacteriological swabs
Contamination in the rectal stump after wash-out | during surgery

SECONDARY OUTCOMES:
septic complications | within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baselland Bruderholz, Bruderholz, Switzerland